CLINICAL TRIAL: NCT04027491
Title: Innovative Low-cost Solutions Based on Virtual Reality for Upper Limb Home-based Rehabilitation in Multiple Sclerosis
Brief Title: Virtual Reality for Upper Limb Rehabilitation in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cagliari (Other)
Collaborators: Italian Multiple Sclerosis Foundation (Other); Fondazione Don Carlo Gnocchi Onlus (Other); Azienda Sanitaria Locale di Cagliari (Other)
Responsible Party: Principal Investigator, Massimiliano Pau, Associate Professor, Head of the, University of Cagliari
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 102/2018/CE; 2017/R/19 (Other Grant/Funding Number: FISM)
Record Dates: First submitted 2019-07-16; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis
Keywords: Rehabilitation; Upper limbs; Virtual Reality
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Interventional, randomized, controlled, cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality intervention (Experimental): Participant undergo 12 treatment sessions, during a 4-week period (3 sessions per week).
  Each intervention session lasts 45 minutes.
  Interventions: Behavioral: Virtual Reality
- Observational (No Intervention): Participant undergo a 4 weeks observational period. No intervention are performed.

INTERVENTIONS:
Behavioral: Virtual Reality — The selected commercial games are aimed mostly to improve upper limb functions. The games will be randomly administered during each session. Each game will be played for approximately 10 minutes, with 5 minutes break between each game session.
  The intervention treatment consists of 12 sessions in 4-week period.
  Arms: Virtual reality intervention

SUMMARY:
This study is aimed to test the efficacy and feasibility of an immersive virtual reality (VR) rehabilitation programs to improve upper-limb motor functions in 24 patients with multiple sclerosis (pwMS), characterized by moderate to severe upper-limb motor dysfunctions. In particular, this study will evaluate the efficacy of VR as novel opportunities to increase treatment engagement and rehabilitation effects.

The effectiveness of the rehabilitation program will be assessed using both clinical tests and state-of-the art motion capture system for human movement analysis.

DETAILED DESCRIPTION:
Recent studies highlighted the high social and economic burden of rehabilitation in multiple sclerosis (MS); in fact its cost is approximately 27% of the overall expenses supported by the national health system. In particular, it has been shown that the physical rehabilitation is effective in treating functional impairments associated to gait, balance and daily life activitites. However, most rehabilitative treatments are performed at hospital or in specialized centers, and this is a factor which strongly reduces the persistence of the positive effects in the long-term.

In this context, it appears important to highlight that rehabilitative treatments are often focused on lower limbs functional impairments, while upper limbs dysfunctions seem less considered although approximately 50% of pwMS complain about issues like reduction of manual dexterity and fine motor abilities as well as movements' slowness. Moreover, significantly lower is also the number of the studies focused on upper limbs rehabilitation, if compared to those about walking or balance and also if compared with upper limbs studies in other neurologic diseases like stroke.

A support in overcoming such issues might be provided by the adoption of low-cost devices originally designed for entertainment purposes (e.g. Nintendo Wii or Microsoft Kinect) which have been shown effective in improving some aspects of disability. Nevertheless, while rehabilitation protocols which make use of such system often relies on software designed for healthy individuals, it should be essential to have available routines specifically designed for the MS needs.

On the basis of these considerations, this project intends to design, develop and test an innovative low-cost hardware/software platform for home-based upper limbs rehabilitation based on virtual reality.

In particular, the software will reproduce scenarios of actual daily living activities with increasing complexity to ensure a good degree of transferability of the training into real life.

The strength of this approach lies basically on three factors:

1. Use of commercial low-cost VR systems (e.g. Oculus Rift)
2. Use of public domain software for the Virtual Reality package (i.e. Unity 3D)
3. Availability of kinematic data derived from the analysis of the hand trajectories, which allow clinicians to characterize the performance of the participants as well as his/her progresses The effectiveness of the platform will be tested in laboratory using state-of-the-art motion capture system for human movement analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Definite MS diagnosis, sub-type Relapsing-Remitting or Secondary Progressive
* Clinically stable
* No relapses at the time of the enrolment in the study
* Able to understand the informed consent process and provide consent to participate in the study
* 9-Hole Peg Test score > 30 seconds

Exclusion Criteria:

* Relapses occurring over the past 3 months
* History of seizures
* Severe blurred vision
* Concomitant auditory and vestibular deficits
* Presence of other neurological, orthopaedic (non-MS related), psychiatric or cognitive impairments that would interfere with the execution of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-06-03 (Estimated); Study Completion 2022-06-03 (Estimated)

PRIMARY OUTCOMES:
Change in box and block score | Baseline (T0), immediately after the end of the treatment (+4 weeks, T1), +8 weeks from the baseline (T2)
  The Box and Block Test measures unilateral gross manual dexterity. Score consists of the number of blocks transferred from one compartment to the other compartment in 60 seconds (score each hand separately). Higher values indicate better performance.
  Reference value for unaffected population is 55 blocks/min.

SECONDARY OUTCOMES:
Change in Nine-Hole Peg score | Baseline (T0), immediately after the end of the treatment (+4 weeks, T1), +8 weeks from the baseline (T2)
  The Nine-Hole Peg Test measures finger dexterity. Score consists of the time to place and remove one by one the holes on the board, as quickly as possible. Higher values indicate worse performance.

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Pau, PhD, Principal Investigator — University of Cagliari
Locations (1):
- Laboratorio di Biomeccanica ed Ergonomia industriale - Università degli Studi di Cagliari, Monserrato, Cagliari, Italy